CLINICAL TRIAL: NCT02109562
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy, Safety and Tolerability of RBP-7000 as a Treatment in Subjects With Acute Schizophrenia Over 8 Weeks (2 Subcutaneous Doses)
Brief Title: Randomized, Double-blind, Placebo Controlled, Multi-center and Tolerability of RBP-7000 in Schizophrenia Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RB-US-09-0010
Record Dates: First submitted 2014-03-19; First posted 2014-04-10 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Schizophrenic; Schizophrenias; Risperidone
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- RBP-7000 90 mg (Experimental): Risperidone tablets given during the screening period to check for sensitivity. RBP-7000 administered as a 90 mg subcutaneous injection on Days 1 and 29 for a total of two injections.
  Interventions: Drug: RBP-7000; Drug: Risperidone
- RBP-7000 120 mg (Experimental): Risperidone tablets given during the screening period to check for sensitivity. RBP-7000 administered as a 120 mg subcutaneous injection on Days 1 and 29 for a total of two injections.
  Interventions: Drug: RBP-7000; Drug: Risperidone
- Placebo (Placebo Comparator): Risperidone tablets given during the screening period to check for sensitivity. Placebo administered by subcutaneous injection on Days 1 and 29 for a total of two injections.
  Interventions: Drug: Placebo; Drug: Risperidone

INTERVENTIONS:
Drug: RBP-7000 — RBP-7000 90 mg and 120 mg were a mixture of the ATRIGEL Delivery System and 90 mg and 120 mg risperidone, respectively. The ATRIGEL Delivery System allows for sustained-release of risperidone in a controlled manner. Subcutaneous RBP-7000 injections on Days 1 and 29 in the lower quadrant of the abdomen rotating right and left on day 1 and 29.
  Other Names: risperidone in Atrigel
  Arms: RBP-7000 120 mg; RBP-7000 90 mg
Drug: Placebo — Subcutaneous injection of placebo using the ATRIGEL Delivery System on Days 1 and 29 in the lower quadrant of the abdomen rotating right and left on day 1 and 29.
  Arms: Placebo
Drug: Risperidone — Oral risperidone 0.25 mg tablets daily for the first two days of the screening period. The two 0.25 mg tablets confirmed whether study participants had any negative reaction to risperidone prior to receiving a long-acting injection of risperidone (RBP-7000).
  Other Names: Risperdal

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of RBP-7000 compared with placebo in the treatment of patients with schizophrenia.

This will be a double-blind, placebo-controlled, Phase III study with 90 mg and 120 mg doses of RBP-7000 compared with placebo over an 8-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18 to 55 years, inclusive
* Diagnosis of schizophrenia as defined by Diagnostic and Statistical Manual, Edition 4, text revision (DSM-IV-TR) criteria
* Subjects who are deemed "valid" by the State, Assessability, Face, Ecological, and Rule (SAFER) interview
* Subjects who are otherwise healthy on the basis of their physical examination

Exclusion Criteria:

* Subjects who have an improvement in their total Positive and Negative Syndrome Scale (PANSS) score of 20% or greater between the initial screening visit and the first day of treatment.
* Subjects taking daily oral risperidone at a dose ≥ 6 mg/day
* Subjects who have received a depot antipsychotic within 120 days of screen
* Subjects with treatment resistant schizophrenia, as judged by the investigator, who have been treated with antipsychotics for adequate durations and with adequate dosages.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 354 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Developoment Manager, Study Director — Indivior Inc.
Locations (32):
- United States (32):
  - Woodland International Research Group, Inc., Little Rock, Arkansas
  - Woodland International Research Group, Inc., Springdale, Arkansas
  - Comprehensive Clinical Development - Cerritos, CA, Cerritos, California
  - Synergy Clinical Research of Escondido, Escondido, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Collaborative Neuroscience Networks, Inc., Long Beach, California
  - Apostle Clinical Trials, Inc., Long Beach, California
  - Pacific Research Partners, Oakland, California
  - Excell Research, Inc., Oceanside, California
  - CNRI- Los Angeles, LLC, Pico Rivera, California
  - CNRI - San Diego, LLC, San Diego, California
  - Innovative Clinical Research, Fort Lauderdale, Florida
  - Behavioral Clinical Research, Inc., North Miami, Florida
  - Florida Clinical Research Center, LLC, Orlando, Florida
  - Uptown Research Institute, Chicago, Illinois
  - Alexian Brothers Behavioral Health Hospital, Hoffman Estates, Illinois
  - Via Christi Research, Wichita, Kansas
  - Lake Charles Clinical Trials, LLC, Lake Charles, Louisiana
  - J. Gary Booker, MD, APMC, Shreveport, Louisiana
  - St. Louis Clinical Trials, St Louis, Missouri
  - PsychCare Consultants Research, St Louis, Missouri
  - Altea Research Institute, Las Vegas, Nevada
  - CRI Lifetree, Marlton, New Jersey
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - Midwest Clinical Research Center, LLC, Dayton, Ohio
  - Oklahoma Clinical Research Center, Oklahoma City, Oklahoma
  - CRI Lifetree, Philadelphia, Pennsylvania
  - FutureSearch Clinical Trials, L.P., Austin, Texas
  - Community Clinical Research, Inc., Austin, Texas
  - FutureSearch Clinical Trials, L.P., Dallas, Texas
  - Pillar Clinic Research, LLC, Dallas, Texas

REFERENCES:
- [Derived] Andrade C. Prazosin for Alcohol Use Disorder: Reply to Sinha. J Clin Psychiatry. 2021 Sep 21;82(6):21lr14076a. doi: 10.4088/JCP.21lr14076a. No abstract available. PMID 34551220
- [Derived] Sinha R. Prazosin for Alcohol Use Disorder: A Clarification. J Clin Psychiatry. 2021 Sep 21;82(6):21lr14076. doi: 10.4088/JCP.21lr14076. No abstract available. PMID 34551219
- [Derived] Le Moigne A, Csernansky J, Leadbetter RA, Andorn AC, Graham JA, Heath AT, Walling DP, Newcomer JW, Marder SR. PANSS Individual Item and Marder Dimension Analyses From a Pivotal Trial of RBP-7000 (Monthly Extended-Release Risperidone) in Schizophrenia Patients. J Clin Psychiatry. 2021 Sep 21;82(5):21m13906. doi: 10.4088/JCP.21m13906. PMID 34551218

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 538 subjects were screened for study participation at 33 sites in the US, including 354 subjects randomly assigned to treatment. Four subjects were found to be randomized incorrectly; therefore, they were withdrawn from the study and did not receive study drug (counted as 'Physician Decision' for reason d/c below).
Period: Overall Study
Arm/Group | RBP-7000 90 mg | RBP-7000 120 mg | Placebo
Started | 116 | 119 | 119
Safety (Randomized and received at least one dose of study drug) | 115 | 117 | 118
Intent to Treat (ITT) (Randomized, dosed, had a baseline and 1 or more post baseline efficacy measurements.) | 111 | 114 | 112
Completed | 90 | 85 | 84
Not Completed | 26 | 34 | 35
Not completed — Insufficient clinical response | 2 | 0 | 4
Not completed — Adverse Event | 0 | 2 | 3
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 3 | 1
Not completed — Withdrawal by Subject | 20 | 25 | 21
Not completed — Physician Decision | 3 | 4 | 5

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | RBP-7000 90 mg | RBP-7000 120 mg | Placebo | Total
Number analyzed (Participants) | 115 | 117 | 118 | 350
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (9.41) | 40.6 (9.45) | 42.4 (9.07) | 41.1 (9.33)
Age, Customized [Count of Participants; unit: Participants]
  20 years and under | 1 | 2 | 1 | 4
  21 to 30 years | 16 | 20 | 16 | 52
  31 to 40 years | 38 | 32 | 28 | 98
  41 to 50 years | 41 | 43 | 49 | 133
  51 to 55 years | 19 | 20 | 24 | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 31 | 31 | 82
  Male | 95 | 86 | 87 | 268
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 10 | 26
  Not Hispanic or Latino | 108 | 107 | 107 | 322
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    White | 28 | 30 | 27 | 85
    Black or African American | 83 | 83 | 88 | 254
    Asian | 1 | 3 | 1 | 5
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 3
    Other | 2 | 0 | 1 | 3
Weight [Mean (Standard Deviation); unit: kg] | 90.60 (18.895) | 89.01 (20.462) | 91.84 (22.885) | 90.49 (20.802)
Height [Mean (Standard Deviation); unit: cm] | 175.1 (9.09) | 174.3 (9.95) | 173.1 (10.91) | 174.1 (10.02)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.576 (5.938) | 29.376 (6.664) | 30.706 (7.293) | 29.890 (6.667)
Waist-to-Hip Ratio [Mean (Standard Deviation); unit: ratio] — A measurement of abdominal fat.
  ratio | 0.947 (0.078) | 0.936 (0.072) | 0.944 (0.090) | 0.942 (0.080)
Previous Antipsychotic Treatment [Count of Participants; unit: Participants]
  Yes | 114 | 116 | 118 | 348
  No | 1 | 1 | 0 | 2
Age at First Schizophrenia Diagnosis [Mean (Standard Deviation); unit: years] | 25.5 (8.21) | 26.9 (8.48) | 26.6 (9.25) | 26.3 (8.66)

OUTCOME MEASURES:

1. Primary Outcome: Mixed Model for Repeated Measures (MMRM) Analysis of Change From Baseline to End of Treatment in the Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor judgement, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score is the sum of all 30 PANSS items and ranges from 30 to 210, with 30 indicating absence of symptoms of schizophrenia and 210 indicating extreme ratings of all 30 symptoms. Negative change from baseline scores indicate improvements in symptoms.
  Estimates (least square means and standard errors), 2-sided confidence intervals, and -1-sided P values are based on a repeated-measures linear regression model of the change from baseline score, with fixed effects for visit as a categorical variable, baseline score, treatment and treatment by visit interaction, assuming an unstructured covariance matrix.
Time Frame: Day 1 prior to treatment (Baseline), Days 15, 29, 43 and 57 or early discontinuation
Population: Intent to treat (ITT) population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | RBP-7000 90 mg | RBP-7000 120 mg | Placebo
Number analyzed (Participants) | 111 | 114 | 112
units on a scale | -15.367 (1.2230) | -16.456 (1.2073) | -9.219 (1.2162)
Statistical Analysis 1: Comparison: RBP-7000 90 mg vs Placebo; Estimates, standard errors (SE), 2-sided confidence intervals (CIs), and -1-sided P values are based on a repeated-measures linear regression model of the change from baseline score, with fixed effects for visit as a categorical variable, baseline score, treatment and treatment by visit interaction, assuming an unstructured covariance matrix; Test type: Superiority; p = 0.0004, repeated measure linear regression model — For evaluation of treatment differences, compare against a 1-sided adjusted P value with significance at <0.025. The P values have been adjusted for multiple comparisons using Dunnett's procedure; Mean Difference (Final Values) = -6.148, 95% CI 2-sided [-9.982 to -2.314], Standard Error of Mean 1.7261 — RBP-7000 90 mg - Placebo
Statistical Analysis 2: Comparison: RBP-7000 120 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, repeated measure linear regression model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.237, 95% CI 2-sided [-11.045 to -3.429], Standard Error of Mean 1.7141 — RBP-7000 120 mg - Placebo

2. Secondary Outcome: Mixed Model for Repeated Measures (MMRM) Analysis of Change From Baseline to End of Treatment in Clinical Global Impression - Severity Scale (CGI-S)
Description: The CGI-S rating scale is a 7-point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Negative change from baseline scores indicate improvement in the severity of illness.
  Estimates (least square means and standard errors), 2-sided confidence intervals, and -1-sided P values are based on a repeated-measures linear regression model of the change from baseline score, with fixed effects for visit as a categorical variable, baseline score, treatment and treatment by visit interaction, assuming an unstructured covariance matrix.
Time Frame: Day 1 prior to treatment (Baseline), Days 15, 29, 43 and 57 or early discontinuation
Population: Intent to treat population (ITT)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | RBP-7000 90 mg | RBP-7000 120 mg | Placebo
Number analyzed (Participants) | 111 | 114 | 112
units on a scale | -0.868 (0.0662) | -0.914 (0.0654) | -0.518 (0.0659)
Statistical Analysis 1: Comparison: RBP-7000 90 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0002, repeated measure linear regression model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.350, 95% CI 2-sided [-0.557 to -0.143], Standard Error of Mean 0.0934 — RBP-7000 90 mg - Placebo
Statistical Analysis 2: Comparison: RBP-7000 120 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, repeated measure linear regression model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.396, 95% CI 2-sided [-0.602 to -0.190], Standard Error of Mean 0.0928 — RBP-7000 120 mg - Placebo

3. Secondary Outcome: Summary of Participants With Treatment-Emergent Adverse Events (TEAE)
Description: An adverse event (AE) is defined as any study-related event that represents a change (positive or negative) in frequency or severity from a baseline (prestudy) event (if any), regardless of the presence of causal relationship or medical significance. Treatment-emergent adverse events are defined as any adverse event with a start date on or after the first study dose date. AEs are determined by the Investigator to be related or not related to the study drug.
  A serious AE (SAE) is defined by federal regulation as any AE occurring at any dose that results in any of the following outcomes: death, life-threatening AE, hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity, or a congenital anomaly/birth defect. Although a subject may have had 2 or more adverse experiences the subject is counted only once in a category. The same subject may appear in different categories.
Time Frame: Day 1 to Week 8
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | RBP-7000 90 mg | RBP-7000 120 mg | Placebo
Number analyzed (Participants) | 115 | 117 | 118
Participants
  No TEAEs | 34 | 26 | 37
  1 or more TEAEs | 81 | 91 | 81
  Related TEAE | 58 | 65 | 50
  Serious TEAE | 0 | 1 | 1
  Serious, related TEAE | 0 | 0 | 0
  TEAE causing discontinuation | 0 | 2 | 3
  Death | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Week 8
Arm/Group | RBP-7000 90 mg | RBP-7000 120 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/117 | 0/118
Serious Adverse Events (participants affected / at risk) | 0/115 | 1/117 | 1/118
Other Adverse Events (participants affected / at risk) | 65/115 | 70/117 | 64/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RBP-7000 90 mg (N=115) | RBP-7000 120 mg (N=117) | Placebo (N=118)
Chest pain (General disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RBP-7000 90 mg (N=115) | RBP-7000 120 mg (N=117) | Placebo (N=118)
Injection site pain (General disorders) | 18 | 26 | 23
Headache (Nervous system disorders) | 20 | 18 | 28
Weight increased (Investigations) | 15 | 15 | 4
Constipation (Gastrointestinal disorders) | 8 | 9 | 6
Toothache (Gastrointestinal disorders) | 9 | 8 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 8 | 5
Injection site erythema (General disorders) | 7 | 5 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 6 | 3
Akathisia (Nervous system disorders) | 3 | 8 | 5
Anxiety (Psychiatric disorders) | 3 | 8 | 6
Dyspepsia (Gastrointestinal disorders) | 4 | 7 | 11
Nausea (Gastrointestinal disorders) | 5 | 6 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 5 | 9
Somnolence (Nervous system disorders) | 6 | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 9 | 6
Insomnia (Psychiatric disorders) | 4 | 3 | 7
Nodule (General disorders) | 3 | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Proposed publications shall be submitted to Sponsor 30 days prior to submission for publication, and may be withheld for an additional period, up to 90 days, to allow Sponsor to file patent applications. If a multicenter publication isn't submitted for publication within 12 months of the conclusion of the Study at all sites, or is published in a shorter period, the results from the institution's site may be published individually.